CLINICAL TRIAL: NCT02413892
Title: Impact of a Loading Dose of Caspofungin on Pharmacokinetic and Pharmacodynamic Parameters Target Achievements for Severe Candida Infections in ICU Patients
Brief Title: Impact of a Loading Dose of Caspofungin in Invasive Candidiasis in ICU Patients
Acronym: CASPOLOAD
Status: Completed | Type: Observational
Sponsor: Outcome Rea (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: OCR001
Record Dates: First submitted 2015-03-09; First posted 2015-04-10 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2016-04

CONDITIONS: Candida Infections
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The samples were collected as part of patient care in medical monitoring and resuscitation infectious Bichat Hospital. They will be used to search within the site.
  In these severe patients, arterial catheter is systematically implemented. The investigators plan to collect thru this catheter five blood 4ml tubes on 24hours to measure the pharmacodynamic parameters of caspofungin.
Oversight: Data Monitoring Committee: No

SUMMARY:
Echinocandins are the drug of choice in severe candida infections. Efficacy of echinocandins is related to concentration and area under the curve (AUC) of the drug.

Available pharmacokinetic studies found that concentration of echinocandins mainly caspofungin is sub-optimal in severe candida infections in intensive care unit (ICU) patients.

Higher dose of caspofungin has been proven to be safe in critically ill patients but its impact on the ability to reach PK/PD target is unknown.

The aim of this study is to evaluate the impact of a loading dose of caspofungin on PK/PD parameters within the first 24-hours.

DETAILED DESCRIPTION:
Invasive fungal infections are associated to a high mortality rate in ICU, partly because of a delayed treatment.

PK/PD targets for caspofungin are the peak concentration over minimal inhibitory concentration (MIC) ratio which should reach 10 and the area under the inhibitory curve (AUIC) which should be over 200. High distribution volume in ICU patients and increase of MICs due to extensive use of antifungal agents make optimal concentration difficult to obtain. High doses up to 150mg of caspofungin have been reported to be safe. Thus, in our unit, a loading dose of 140mg of caspofungin is a standard practice but was never rigorously evaluated.

The aim of the present study is to measure the impact of a loading dose of 140mg of caspofungin on the pharmacokinetic parameters in the first 24 hours of treatment.

The AUIC and maximal concentration (CMax) / (MIC) according to the recovered yeasts will be measured. The investigators also planned a Monte-Carlo simulation using MICs obtained from clinically relevant candida strains isolated in Bichat and Grenoble hospitals in order to evaluate the percentage of patients appropriately treated within the first 24 hours according to Candida species and previous use of antifungals.

Recovered strains from epidemiological studies will be used for PKPD modelling and will use s. A second Monte-Carlo simulation will be done using data from the Amarcand 2 study.

All MICs will be determined using E-test ( Biomerieux® KIT's) without specifying any breakpoints as MICs and not breakpoints per se will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in intensive care
* Age> 18 years
* Patient with a central catheter
* Patient with invasive mechanical ventilation
* Patient receiving more than 0.1 mcg / kg / min of adrenaline or noradrenaline
* Patient treated for proven (positive blood cultures or positive specimen obtained during a surgical or percutaneous puncture) or suspected (risk factor, extra digestive colonization, absence of other uncontrolled bacterial infections, candida score> 3) invasive candidiasis.
* Patient affiliated to medical insurance

Exclusion Criteria:

* Expected length of stay under 48H
* Age <18 years
* Pregnant or breastfeeding women
* Limited or sustained life support therapy
* Patient unable to legally consent
* History of Allergy, hypersensitivity or intolerance to echinocandins or Drug excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients for whom the decision to start antifungal therapy with caspofungin loading dose was taken
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Area Under the inhibitory curve (AUIC) | 24 hours after the loading dose
  Six samples (before infusion; 2, 3, 5, 7 and 24 hours after infusion) will be obtained between inclusion and 24 hours to calculate the area under the curve. MIC will be determined with E-test technique.

SECONDARY OUTCOMES:
Peak concentration over MIC (Cmax/MIC) | 2 hours avec the loading dose
  One blood sample will be obtained. MIC will be determined with E-test technique.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois TIMSIT, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Reanimation Medicale et Infectieuse-Hopital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shields RK, Nguyen MH, Press EG, Updike CL, Clancy CJ. Caspofungin MICs correlate with treatment outcomes among patients with Candida glabrata invasive candidiasis and prior echinocandin exposure. Antimicrob Agents Chemother. 2013 Aug;57(8):3528-35. doi: 10.1128/AAC.00136-13. Epub 2013 May 13. PMID 23669387
- [Background] Safdar A, Rodriguez G, Rolston KV, O'Brien S, Khouri IF, Shpall EJ, Keating MJ, Kantarjian HM, Champlin RE, Raad II, Kontoyiannis DP. High-dose caspofungin combination antifungal therapy in patients with hematologic malignancies and hematopoietic stem cell transplantation. Bone Marrow Transplant. 2007 Feb;39(3):157-64. doi: 10.1038/sj.bmt.1705559. PMID 17245424
- [Background] Betts RF, Nucci M, Talwar D, Gareca M, Queiroz-Telles F, Bedimo RJ, Herbrecht R, Ruiz-Palacios G, Young JA, Baddley JW, Strohmaier KM, Tucker KA, Taylor AF, Kartsonis NA; Caspofungin High-Dose Study Group. A Multicenter, double-blind trial of a high-dose caspofungin treatment regimen versus a standard caspofungin treatment regimen for adult patients with invasive candidiasis. Clin Infect Dis. 2009 Jun 15;48(12):1676-84. doi: 10.1086/598933. PMID 19419331
- [Background] Louie A, Deziel M, Liu W, Drusano MF, Gumbo T, Drusano GL. Pharmacodynamics of caspofungin in a murine model of systemic candidiasis: importance of persistence of caspofungin in tissues to understanding drug activity. Antimicrob Agents Chemother. 2005 Dec;49(12):5058-68. doi: 10.1128/AAC.49.12.5058-5068.2005. PMID 16304173
- [Background] Sinnollareddy M, Peake SL, Roberts MS, Lipman J, Roberts JA. Using pharmacokinetics and pharmacodynamics to optimise dosing of antifungal agents in critically ill patients: a systematic review. Int J Antimicrob Agents. 2012 Jan;39(1):1-10. doi: 10.1016/j.ijantimicag.2011.07.013. Epub 2011 Sep 16. PMID 21925845
- [Background] Nguyen TH, Hoppe-Tichy T, Geiss HK, Rastall AC, Swoboda S, Schmidt J, Weigand MA. Factors influencing caspofungin plasma concentrations in patients of a surgical intensive care unit. J Antimicrob Chemother. 2007 Jul;60(1):100-6. doi: 10.1093/jac/dkm125. Epub 2007 May 24. PMID 17525052
- [Derived] Bailly S, Gautier-Veyret E, Le MP, Bouadma L, Andremont O, Neuville M, Mourvillier B, Sonneville R, Magalhaes E, Lebut J, Radjou A, Smonig R, Wolff M, Massias L, Dupuis C, Timsit JF. Impact of Loading Dose of Caspofungin in Pharmacokinetic-Pharmacodynamic Target Attainment for Severe Candidiasis Infections in Patients in Intensive Care Units: the CASPOLOAD Study. Antimicrob Agents Chemother. 2020 Nov 17;64(12):e01545-20. doi: 10.1128/AAC.01545-20. Print 2020 Nov 17. PMID 32958709